CLINICAL TRIAL: NCT00612352
Title: Intravenous Alcohol Administration Using BrAc Method in Healthy Subjects With and Without a Family History of Alcoholism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 0304025194; VA Alcohol Research Center (Other Grant/Funding Number: VA Alcohol Research Center Grant); P50AA012870 (NIH)
Record Dates: First submitted 2007-12-27; First posted 2008-02-11 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family HIstory Positive (Active Comparator): Subjects with a positive family history of alcoholism.
  Interventions: Drug: Ethanol High Dose, Ethanol Low Dose, and Placebo
- Family History Negative (Active Comparator): Subjects with a negative family history of alcoholism.
  Interventions: Drug: Ethanol High Dose, Ethanol Low Dose, and Placebo

INTERVENTIONS:
Drug: Ethanol High Dose, Ethanol Low Dose, and Placebo — Three test days will involve administration of placebo, ethanol high dose (BrAc=100mg%) or ethanol low dose (BrAc=40mg%)intravenously for approximately 20 minutes, until the target BrAc is achieved. Once BrAc is achieved (40mg% or 100mg%) it will be maintained using a clamp procedure for 60 minutes.
  Other Names: intravenous

SUMMARY:
The proposed study is the first to explore the contribution of brain glutamate systems, a major target of ethanol in the brain, to the vulnerability to develop alcoholism. This study may lead to an enhanced understanding of the underlying neurobiological mechanism in high risk individuals that may lead to the transition from moderate to excessive use of alcohol.

DETAILED DESCRIPTION:
Males and females with a paternal family history of alcoholism have a high risk for developing alcoholism. These individuals have been shown to have decreased dysphoric responses to alcohol self-administration that may promote the excessive use of alcohol. Ethanol has been shown to be an antagonist at the N-methyl-D-aspartate (NMDA) glutamate receptor. We have recently shown that sober alcoholics have decreased dysphoric response to the NMDA antagonist, ketamine. We propose to test the hypothesis that this characteristic exists as a vulnerability factor in those individuals susceptible to develop alcoholism. Specifically, the objective is to determine whether individuals with a family history positive (FHP) for alcoholism will experience less dysphoric, anxiogenic, and psychotogenic effects to alcohol infusion when compared to family history negative (FHN) control subjects.

Male and female subjects, FHP (biological father and one other first degree relative) between the ages of 21-30, and matched controls (FHN) will complete 3 test days in a randomized balanced order under double-blind conditions. Test days will involve administration of placebo or one of two ethanol doses (target BrAc=40mg%, or target BrAc=100mg%) intravenously for 20 minutes, until the target BrAc is achieved. Once BrAc is achieved (40mg% or 100mg%) it will be maintained using a clamp procedure for over 60 minutes. Outcome measures include the Positive and Negative Symptom Scale, visual analog scales of mood state, (i.e. anxiety) and the Clinician-Administered Dissociative States Scale (CADSS) to measure perceptual responses to alcohol. Secondary measures include visual analog scales for high, similarity to ethanol, Mini Mental Status Examination (MMSE), Placement of electrodes, Biphasic Alcohol Effects Scale, Hopkins Verbal Learning, and number of drinks scale, aspects of craving for alcohol and tests of cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female between the ages of 21 and 30 years;
2. medically and neurologically healthy on the basis of history, physical examination, EKG, Screening laboratories absence of current and/or past substance abuse on the basis of history and urine toxicology and breath alcohol levels at screening and on each test day.

For Family History Positive (FHP) Subjects: 1) Biological father and another first or second-degree biological relative with history of alcoholism by Family History Assessment Module (FHAM) developed by COGA.

Exclusion Criteria:

1. DSM-IV psychiatric and substance abuse (excluding alcohol abuse) diagnosis by history on psychiatric evaluation that includes a structured diagnostic interview (Structured Clinical Interview for Diagnostic and Statistical Manual (DSM)-IV Axis I Disorders (SCID))
2. Subjects who meet criteria for alcohol abuse and express an interest in stopping alcohol use and/or express an interest in treatment or are currently enrolled in treatment for alcoholism, or have sought treatment in the last 6 months.
3. history of counseling or psychotherapy; except family therapy centered around another family member
4. extended unwillingness to remain alcohol-free for 48 hours prior to test days;
5. for women: positive pregnancy test at screening or intention to engage in unprotected sex during the study
6. alcohol naïve
7. Adoptee and no contact with family members.

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2001-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ismene L Petrakis, MD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Result] Ralevski E, Perrino A, Acampora G, Koretski J, Limoncelli D, Petrakis I. Analgesic effects of ethanol are influenced by family history of alcoholism and neuroticism. Alcohol Clin Exp Res. 2010 Aug;34(8):1433-41. doi: 10.1111/j.1530-0277.2010.01228.x. Epub 2010 May 21. PMID 20497133
- [Result] Perrino AC Jr, Ralevski E, Acampora G, Edgecombe J, Limoncelli D, Petrakis IL. Ethanol and pain sensitivity: effects in healthy subjects using an acute pain paradigm. Alcohol Clin Exp Res. 2008 Jun;32(6):952-8. doi: 10.1111/j.1530-0277.2008.00653.x. Epub 2008 Apr 26. PMID 18445106

RESULTS

PARTICIPANT FLOW:
Groups:
- Family History Negative: Subjects with no family history of alcoholism.
Period: Overall Study
Arm/Group | Family History Positive | Family History Negative
Started | 65 | 115
40%mg & 100%mg (Subjects that completed 2 test days (40%mg ethanol & 100%mg ethanol)) | 1 | 1
Placebo & 100%mg (Subjects that completed 2 test days (placebo & 100%mg ethanol)) | 1 | 0
100%mg (Subjects that completed 1 test day (100%mg ethanol)) | 2 | 1
40%mg (Subjects that completed 1 test day (40%mg ethanol)) | 1 | 0
Placebo (Subjects that completed 1 test day (placebo)) | 4 | 4
Completed (Completed all three test dates.) | 56 | 109
Not Completed | 9 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 3 | 5
Not completed — moved out of state | 1 | 0
Not completed — didn't return calls/show up on test date | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Family History Positive | Family History Negative | Total
Number analyzed (Participants) | 65 | 115 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.06 (2.97) | 24.1 (2.38) | 24.08 (2.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 56 | 88
  Male | 33 | 59 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 14 | 24
  White | 51 | 88 | 139
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 13 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinks Felt Consumed at Baseline
Description: The Number of Drinks Scale asks Subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: drinks felt consumed
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
drinks felt consumed
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0 (0) | 0 (0)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 108
  Alcohol 40mg% | 0 (0) | 0 (0)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 109
  Alcohol 100mg% | 0 (0) | 0.04 (0.23)

2. Primary Outcome: Number of Drinks Felt Consumed at 10 Minutes
Description: The Number of Drinks Scale asks Subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: 10 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: drinks felt consumed
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
drinks felt consumed
  Placebo: number analyzed (Participants) | 56 | 92
  Placebo | 0.07 (0.42) | 0.08 (0.37)
  Alcohol 40mg%: number analyzed (Participants) | 53 | 90
  Alcohol 40mg% | 0.49 (0.8) | 0.7 (0.92)
  Alcohol 100mg%: number analyzed (Participants) | 53 | 91
  Alcohol 100mg% | 0.76 (1.07) | 1.15 (1.18)

3. Primary Outcome: Number of Drinks Felt Consumed at 30 Minutes
Description: The Number of Drinks Scale asks Subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: 30 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: drinks felt consumed
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
drinks felt consumed
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.2 (0.5) | 0.27 (0.67)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 1.88 (1.11) | 2.03 (1.68)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 110
  Alcohol 100mg% | 3.65 (1.61) | 3.86 (2.0)

4. Primary Outcome: Number of Drinks Felt Consumed at 110 Minutes
Description: The Number of Drinks Scale asks Subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: 110 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: drinks felt consumed
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
drinks felt consumed
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.1 (0.4) | 0.09 (0.4)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 108
  Alcohol 40mg% | 0.97 (0.97) | 1.2 (1.39)
  Alcohol 100mg%: number analyzed (Participants) | 58 | 109
  Alcohol 100mg% | 3.22 (1.61) | 3.64 (2.0)

5. Primary Outcome: Number of Drinks Felt Consumed at 140 Minutes
Description: The Number of Drinks Scale asks Subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: 140 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: drinks felt consumed
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
drinks felt consumed
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.03 (0.18) | 0.04 (0.23)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0.33 (0.63) | 0.46 (0.88)
  Alcohol 100mg%: number analyzed (Participants) | 58 | 108
  Alcohol 100mg% | 2.12 (1.79) | 2.53 (2.78)

6. Primary Outcome: Number of Drinks Felt Consumed at 170 Minutes
Description: The Number of Drinks Scale asks Subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: 170 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: drinks felt consumed
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
drinks felt consumed
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0 (0) | 0 (0)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0.07 (0.32) | 0.11 (0.39)
  Alcohol 100mg%: number analyzed (Participants) | 59 | 109
  Alcohol 100mg% | 1.19 (1.5) | 1.39 (2.24)

7. Primary Outcome: Number of Drinks Felt Consumed at 230 Minutes
Description: The Number of Drinks Scale asks Subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: 230 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: drinks felt consumed
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
drinks felt consumed
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0 (0) | 0 (0)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0.03 (0.26) | 0.03 (0.21)
  Alcohol 100mg%: number analyzed (Participants) | 59 | 110
  Alcohol 100mg% | 0.37 (0.79) | 0.55 (1.16)

8. Primary Outcome: Visual Analog Scale of Similarity to Alcohol - Baseline
Description: Visual Analog Scale of Similarity to Alcohol data using the Likert scale (0 Not at all similar to alcohol - 7 Extremely similar to alcohol) evaluating the similarity of drug effects to alcohol
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.08 (0.64) | 0.13 (0.65)
  Alcohol 40mg%: number analyzed (Participants) | 57 | 109
  Alcohol 40mg% | 0.1 (0.41) | 0.1 (0.62)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 110
  Alcohol 100mg% | 0.02 (0.13) | 0.1 (0.59)

9. Primary Outcome: Visual Analog Scale of Similarity to Alcohol -10 Minutes
Description: as for outcome 8
Time Frame: 10 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 56 | 92
  Placebo | 0.16 (0.73) | 0.12 (0.41)
  Alcohol 40mg%: number analyzed (Participants) | 53 | 90
  Alcohol 40mg% | 0.76 (1.3) | 1.13 (1.6)
  Alcohol 100mg%: number analyzed (Participants) | 53 | 91
  Alcohol 100mg% | 1.59 (2.2) | 1.56 (1.81)

10. Primary Outcome: Visual Analog Scale of Similarity to Alcohol - 30 Minutes
Description: as for outcome 8
Time Frame: 30 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.36 (1.08) | 0.33 (0.69)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 2.05 (2.06) | 2.62 (2.25)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 110
  Alcohol 100mg% | 3.82 (2.05) | 3.98 (1.82)

11. Primary Outcome: Visual Analog Scale of Similarity to Alcohol - 60 Minutes
Description: as for outcome 8
Time Frame: 60 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.36 (1.16) | 0.32 (0.81)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 2.21 (2.27) | 2.52 (2.28)
  Alcohol 100mg%: number analyzed (Participants) | 59 | 107
  Alcohol 100mg% | 3.83 (2.19) | 4.01 (1.98)

12. Primary Outcome: Visual Analog Scale of Similarity to Alcohol - 110 Minutes
Description: as for outcome 8
Time Frame: 110 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.1 (0.4) | 0.14 (0.55)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 1.19 (1.5) | 1.31 (1.73)
  Alcohol 100mg%: number analyzed (Participants) | 58 | 109
  Alcohol 100mg% | 2.97 (2.42) | 3.12 (2.16)

13. Primary Outcome: Visual Analog Scale of Similarity to Alcohol - 140 Minutes
Description: as for outcome 8
Time Frame: 140 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.05 (0.28) | 0.05 (0.35)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0.29 (0.75) | 0.68 (1.31)
  Alcohol 100mg%: number analyzed (Participants) | 58 | 108
  Alcohol 100mg% | 2.29 (2.27) | 2.16 (2.06)

14. Primary Outcome: Visual Analog Scale of Similarity to Alcohol - 170 Minutes
Description: as for outcome 8
Time Frame: 170 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0 (0) | 0.01 (0.09)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0.1 (0.41) | 0.21 (0.63)
  Alcohol 100mg%: number analyzed (Participants) | 59 | 109
  Alcohol 100mg% | 1.37 (1.89) | 1.41 (1.81)

15. Primary Outcome: Visual Analog Scale of Similarity to Alcohol - 230 Minutes
Description: as for outcome 8
Time Frame: 230 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.02 (0.13) | 0 (0)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0.05 (0.29) | 0.05 (0.25)
  Alcohol 100mg%: number analyzed (Participants) | 59 | 110
  Alcohol 100mg% | 0.46 (0.92) | 0.71 (1.42)

16. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedative Baseline
Description: Self-report rating scale used to measure sedative effects (0 not at all sedated - 70 extremely sedated)
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 111
  Placebo | 2.21 (4.47) | 1.8 (3.69)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 1.16 (2.46) | 2.21 (4.68)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 110
  Alcohol 100mg% | 2.02 (4.59) | 2.17 (4.29)

17. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedative - 10 Minutes
Description: Self-report rating scale used to measure sedative effects (0 not at all sedated - 70 extremely sedated)
Time Frame: 10 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 56 | 92
  Placebo | 2.04 (4.11) | 1.85 (3.8)
  Alcohol 40mg%: number analyzed (Participants) | 53 | 90
  Alcohol 40mg% | 1.59 (4.43) | 3.83 (6.91)
  Alcohol 100mg%: number analyzed (Participants) | 53 | 91
  Alcohol 100mg% | 4.3 (8.13) | 4.5 (7.66)

18. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedative - 30 Minutes
Description: Self-report rating scale used to measure sedative effects (0 not at all sedated - 70 extremely sedated)
Time Frame: 30 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 2.1 (4.23) | 2.36 (4.56)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 3.41 (5.26) | 6.16 (9.1)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 109
  Alcohol 100mg% | 7.75 (11.09) | 9.38 (13.75)

19. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedative - 60 Minutes
Description: Self-report rating scale used to measure sedative effects (0 not at all sedated - 70 extremely sedated)
Time Frame: 60 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 111
  Placebo | 2.46 (4.94) | 2.9 (6.35)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 4.17 (6.62) | 6.32 (9.67)
  Alcohol 100mg%: number analyzed (Participants) | 59 | 108
  Alcohol 100mg% | 8.27 (11.55) | 10.45 (14.87)

20. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedative - 110 Minutes
Description: Self-report rating scale used to measure sedative effects (0 not at all sedated - 70 extremely sedated)
Time Frame: 110 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 1.93 (4.11) | 1.92 (5.36)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 4.21 (7.95) | 4.68 (7.38)
  Alcohol 100mg%: number analyzed (Participants) | 58 | 109
  Alcohol 100mg% | 7.5 (10.65) | 9.77 (13.55)

21. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedative - 140 Minutes
Description: Self-report rating scale used to measure sedative effects (0 not at all sedated - 70 extremely sedated)
Time Frame: 140 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 1.34 (3.12) | 1.8 (5.01)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 2.55 (6.55) | 3.39 (6.22)
  Alcohol 100mg%: number analyzed (Participants) | 58 | 108
  Alcohol 100mg% | 6.28 (10.67) | 7.4 (11.88)

22. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedative - 170 Minutes
Description: Self-report rating scale used to measure sedative effects (0 not at all sedated - 70 extremely sedated)
Time Frame: 170 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.79 (2.35) | 1.22 (4.44)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 108
  Alcohol 40mg% | 1.4 (3.98) | 1.96 (4.47)
  Alcohol 100mg%: number analyzed (Participants) | 59 | 109
  Alcohol 100mg% | 3.97 (6.82) | 5.78 (11.52)

23. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedative - 230 Minutes
Description: Self-report rating scale used to measure sedative effects (0 not at all sedated - 70 extremely sedated)
Time Frame: 230 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.62 (2.31) | 1.03 (3.58)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 1.28 (3.38) | 1.56 (4.19)
  Alcohol 100mg%: number analyzed (Participants) | 59 | 110
  Alcohol 100mg% | 2.7 (6.27) | 3.25 (6.15)

24. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulant - Baseline
Description: Self-report rating scale used to measure stimulant effects (0 not at all stimulated - 70 extremely stimulated)
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 3.15 (6.89) | 2.93 (6.6)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 4.59 (9.28) | 4.47 (9.91)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 110
  Alcohol 100mg% | 3.4 (6.73) | 3.55 (7.41)

25. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulant - 10 Minutes
Description: Self-report rating scale used to measure stimulant effects (0 not at all stimulated - 70 extremely stimulated)
Time Frame: 10 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 61 | 115
units on a scale
  Placebo: number analyzed (Participants) | 56 | 92
  Placebo | 3.39 (8.15) | 2.19 (5.7)
  Alcohol 40mg%: number analyzed (Participants) | 53 | 90
  Alcohol 40mg% | 4.23 (9.26) | 3.54 (7.32)
  Alcohol 100mg%: number analyzed (Participants) | 53 | 91
  Alcohol 100mg% | 3.83 (6.34) | 4.19 (7.83)

26. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulant - 30 Minutes
Description: Self-report rating scale used to measure stimulant effects (0 not at all stimulated - 70 extremely stimulated)
Time Frame: 30 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 3.75 (8.31) | 2.79 (6.54)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 5.66 (9.82) | 6.19 (9.28)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 110
  Alcohol 100mg% | 8.97 (12.75) | 10.38 (12.18)

27. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulant - 60 Minutes
Description: Self-report rating scale used to measure stimulant effects (0 not at all stimulated - 70 extremely stimulated)
Time Frame: 60 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 3.75 (8.32) | 2.74 (6.37)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 4.29 (8.61) | 4.82 (8.29)
  Alcohol 100mg%: number analyzed (Participants) | 59 | 108
  Alcohol 100mg% | 7.51 (11.79) | 7.61 (10.32)

28. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulant - 110 Minutes
Description: Self-report rating scale used to measure stimulant effects (0 not at all stimulated - 70 extremely stimulated)
Time Frame: 110 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 3.15 (7.33) | 3.92 (7.39)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 2.83 (7.41) | 3.62 (7.52)
  Alcohol 100mg%: number analyzed (Participants) | 58 | 109
  Alcohol 100mg% | 3 (6.22) | 4.52 (8.06)

29. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulant - 140 Minutes
Description: Self-report rating scale used to measure stimulant effects (0 not at all stimulated - 70 extremely stimulated)
Time Frame: 140 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 3.12 (6.95) | 3.79 (8.56)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 2.79 (6.98) | 3.3 (7.59)
  Alcohol 100mg%: number analyzed (Participants) | 58 | 107
  Alcohol 100mg% | 2.35 (4.66) | 3.79 (7.37)

30. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulant - 170 Minutes
Description: Self-report rating scale used to measure stimulant effects (0 not at all stimulated - 70 extremely stimulated)
Time Frame: 170 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 3.57 (7.82) | 4.1 (8.95)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 108
  Alcohol 40mg% | 2.76 (6.58) | 3.21 (7.47)
  Alcohol 100mg%: number analyzed (Participants) | 59 | 109
  Alcohol 100mg% | 1.63 (3.61) | 3.22 (6.92)

31. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulant - 240 Minutes
Description: Self-report rating scale used to measure stimulant effects (0 not at all stimulated - 70 extremely stimulated)
Time Frame: 240 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 4.77 (10.79) | 3.91 (7.89)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 2.95 (7.08) | 4.27 (9.99)
  Alcohol 100mg%: number analyzed (Participants) | 59 | 110
  Alcohol 100mg% | 1.36 (3.5) | 2.79 (6.46)

32. Secondary Outcome: Visual Analog Scale (VAS) HIGH - Baseline
Description: visual analog scale (VAS): self-report scale used to measure high (0 not at all High - 7 extremely High)
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.08 (0.46) | 0.17 (0.71)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0.09 (0.47) | 0.18 (0.88)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 110
  Alcohol 100mg% | 0.05 (0.29) | 0.11 (0.53)

33. Secondary Outcome: Visual Analog Scale (VAS) HIGH - 10 Minutes
Description: visual analog scale (VAS): self-report scale used to measure high (0 not at all High - 7 extremely High)
Time Frame: 10 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 56 | 92
  Placebo | 0.11 (0.56) | 0.12 (0.47)
  Alcohol 40mg%: number analyzed (Participants) | 53 | 90
  Alcohol 40mg% | 0.25 (0.71) | 0.32 (0.81)
  Alcohol 100mg%: number analyzed (Participants) | 53 | 91
  Alcohol 100mg% | 0.51 (1.01) | 0.52 (1.03)

34. Secondary Outcome: Visual Analog Scale (VAS) HIGH - 30 Minutes
Description: visual analog scale (VAS): self-report scale used to measure high (0 not at all High - 7 extremely High)
Time Frame: 30 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.18 (0.65) | 0.16 (0.55)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0.59 (1.11) | 0.99 (1.51)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 110
  Alcohol 100mg% | 1.83 (2.04) | 1.73 (1.99)

35. Secondary Outcome: Visual Analog Scale (VAS) HIGH - 60 Minutes
Description: visual analog scale (VAS): self-report scale used to measure high (0 not at all High - 7 extremely High)
Time Frame: 60 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.18 (0.85) | 0.19 (0.53)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0.69 (1.33) | 0.9 (1.52)
  Alcohol 100mg%: number analyzed (Participants) | 59 | 107
  Alcohol 100mg% | 1.73 (2.20) | 1.66 (1.96)

36. Secondary Outcome: Visual Analog Scale (VAS) HIGH - 110 Minutes
Description: visual analog scale (VAS): self-report scale used to measure high (0 not at all High - 7 extremely High)
Time Frame: 110 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.05 (0.22) | 0.08 (0.38)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0.29 (0.68) | 0.47 (1.13)
  Alcohol 100mg%: number analyzed (Participants) | 58 | 109
  Alcohol 100mg% | 1.21 (2.02) | 0.96 (1.58)

37. Secondary Outcome: Visual Analog Scale (VAS) HIGH - 140 Minutes
Description: visual analog scale (VAS): self-report scale used to measure high (0 not at all High - 7 extremely High)
Time Frame: 140 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0 (0) | 0.05 (0.3)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0.07 (0.32) | 0.21 (0.77)
  Alcohol 100mg%: number analyzed (Participants) | 58 | 108
  Alcohol 100mg% | 0.85 (1.69) | 0.68 (1.41)

38. Secondary Outcome: Visual Analog Scale (VAS) HIGH - 170 Minutes
Description: visual analog scale (VAS): self-report scale used to measure high (0 not at all High - 7 extremely High)
Time Frame: 170 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.02 (0.13) | 0.04 (0.23)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0.02 (0.13) | 0.06 (0.37)
  Alcohol 100mg%: number analyzed (Participants) | 59 | 109
  Alcohol 100mg% | 0.46 (0.97) | 0.46 (1.13)

39. Secondary Outcome: Visual Analog Scale (VAS) HIGH - 240 Minutes
Description: visual analog scale (VAS): self-report scale used to measure high (0 not at all High - 7 extremely High)
Time Frame: 240 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.02 (0.13) | 0.04 (0.23)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0 (0) | 0.03 (0.29)
  Alcohol 100mg%: number analyzed (Participants) | 59 | 110
  Alcohol 100mg% | 0.05 (0.22) | 0.16 (0.57)

40. Secondary Outcome: Visual Analog Scale (VAS) Drowsy - Baseline
Description: visual analog scale (VAS): self-report scale used to measure Drowsy (0 not at all drowsy - 7 extremely drowsy)
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.61 (1.19) | 0.7 (1.09)
  Alcohol 40mg%: number analyzed (Participants) | 57 | 109
  Alcohol 40mg% | 0.47 (0.89) | 0.71 (1.07)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 110
  Alcohol 100mg% | 0.62 (1.12) | 0.87 (1.32)

41. Secondary Outcome: Visual Analog Scale (VAS) Drowsy - 10 Minutes
Description: visual analog scale (VAS): self-report scale used to measure Drowsy (0 not at all drowsy - 7 extremely drowsy)
Time Frame: 10 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 56 | 92
  Placebo | 0.63 (1.07) | 0.52 (0.94)
  Alcohol 40mg%: number analyzed (Participants) | 53 | 90
  Alcohol 40mg% | 0.47 (0.85) | 0.77 (1.11)
  Alcohol 100mg%: number analyzed (Participants) | 53 | 91
  Alcohol 100mg% | 0.87 (1.13) | 0.96 (1.34)

42. Secondary Outcome: Visual Analog Scale (VAS) Drowsy - 30 Minutes
Description: visual analog scale (VAS): self-report scale used to measure Drowsy (0 not at all drowsy - 7 extremely drowsy)
Time Frame: 30 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.53 (0.99) | 0.51 (0.89)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0.71 (0.99) | 1.03 (1.34)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 110
  Alcohol 100mg% | 1.18 (1.64) | 1.05 (1.75)

43. Secondary Outcome: Visual Analog Scale (VAS) Drowsy - 60 Minutes
Description: visual analog scale (VAS): self-report scale used to measure Drowsy (0 not at all drowsy - 7 extremely drowsy)
Time Frame: 60 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.74 (1.11) | 0.69 (1.24)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 1.03 (1.23) | 1.13 (1.55)
  Alcohol 100mg%: number analyzed (Participants) | 59 | 107
  Alcohol 100mg% | 1.14 (1.71) | 1.27 (1.99)

44. Secondary Outcome: Visual Analog Scale (VAS) Drowsy - 110 Minutes
Description: visual analog scale (VAS): self-report scale used to measure Drowsy (0 not at all drowsy - 7 extremely drowsy)
Time Frame: 110 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.51 (0.92) | 0.56 (1.17)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0.95 (1.32) | 0.98 (1.47)
  Alcohol 100mg%: number analyzed (Participants) | 58 | 109
  Alcohol 100mg% | 1.38 (1.83) | 1.73 (2.16)

45. Secondary Outcome: Visual Analog Scale (VAS) Drowsy - 140 Minutes
Description: visual analog scale (VAS): self-report scale used to measure Drowsy (0 not at all drowsy - 7 extremely drowsy)
Time Frame: 140 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.46 (1.04) | 0.45 (1.04)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0.41 (0.62) | 0.9 (1.46)
  Alcohol 100mg%: number analyzed (Participants) | 58 | 108
  Alcohol 100mg% | 1.35 (1.89) | 1.60 (1.89)

46. Secondary Outcome: Visual Analog Scale (VAS) Drowsy - 170 Minutes
Description: visual analog scale (VAS): self-report scale used to measure Drowsy (0 not at all drowsy - 7 extremely drowsy)
Time Frame: 170 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.16 (0.49) | 0.24 (0.63)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0.26 (0.58) | 0.61 (1.24)
  Alcohol 100mg%: number analyzed (Participants) | 59 | 109
  Alcohol 100mg% | 0.93 (1.48) | 1.16 (1.72)

47. Secondary Outcome: Visual Analog Scale (VAS) Drowsy - 230 Minutes
Description: visual analog scale (VAS): self-report scale used to measure Drowsy (0 not at all drowsy - 7 extremely drowsy)
Time Frame: 230 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 0.15 (0.54) | 0.21 (0.62)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 0.29 (0.77) | 0.35 (0.77)
  Alcohol 100mg%: number analyzed (Participants) | 59 | 110
  Alcohol 100mg% | 0.59 (1.00) | 0.8 (1.16)

48. Secondary Outcome: Hopkins Verbal Learning Task - Immediate Recall - Trial 1
Description: Hopkins Verbal Learning Task (HVLT) - measures verbal memory and hippocampus function. (Three immediate recall trials) (0 no words recalled - 12 all words recalled)
Time Frame: 30 minutes - Trial 1
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 7.26 (1.64) | 7.46 (1.72)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 7.26 (1.32) | 7.17 (1.59)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 110
  Alcohol 100mg% | 6.33 (1.4) | 6.27 (1.63)

49. Secondary Outcome: Hopkins Verbal Learning Task - Immediate Recall - Trial 2
Description: as for outcome 48
Time Frame: 30 minutes - Trial 2
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 9.43 (1.96) | 9.7 (1.86)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 8.95 (1.95) | 9.13 (2.01)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 110
  Alcohol 100mg% | 7.78 (2.02) | 8.11 (2.03)

50. Secondary Outcome: Hopkins Verbal Learning Task - Immediate Recall - Trial 3
Description: as for outcome 48
Time Frame: 30 minutes - Trial 3
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 10.8 (1.4) | 10.69 (1.42)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 10.22 (1.6) | 10.28 (1.71)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 110
  Alcohol 100mg% | 9.05 (1.85) | 8.89 (2.17)

51. Secondary Outcome: Hopkins Verbal Learning Task - Delay Recall
Description: Hopkins Verbal Learning Task (HVLT) - measures verbal memory and hippocampus function. (Delay Recall: 30 minutes after Trials 1-3 were given) (0 no words recalled - 12 all words recalled)
Time Frame: 60 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
units on a scale
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 10.48 (1.82) | 10.08 (2.11)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 9.41 (2.15) | 9.43 (2.21)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 108
  Alcohol 100mg% | 7.08 (2.81) | 6.796 (2.95)

52. Secondary Outcome: Pegboard Task - Baseline (Dominant Hand)
Description: The pegboard task is a measure of coordination that measures reaction time; how long a subject takes to insert pegs into a pegboard puzzle, first using their dominant hand then using their non-dominant hand. A quicker time indicates greater coordination. Scores are timed in seconds
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
seconds
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 63.64 (8.58) | 61.58 (9.95)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 63.12 (9.38) | 62.4 (9.23)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 110
  Alcohol 100mg% | 64.07 (9.27) | 63.4 (21.4)

53. Secondary Outcome: Pegboard Task - 30 Minutes (Dominant Hand)
Description: as for outcome 52
Time Frame: 30 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
seconds
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 68.32 (11.74) | 65.05 (11.37)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 67.12 (11.69) | 67.26 (14.46)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 110
  Alcohol 100mg% | 76.92 (12.64) | 76.74 (16.43)

54. Secondary Outcome: Pegboard Task - Baseline (Non-Dominant Hand)
Description: as for outcome 52
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
seconds
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 69.36 (11.03) | 66.85 (10.03)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 70.19 (11) | 67.87 (10.28)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 110
  Alcohol 100mg% | 70.66 (10.38) | 67.16 (11.03)

55. Secondary Outcome: Pegboard Task - 30 Minuites (Non-Dominant Hand)
Description: as for outcome 52
Time Frame: 30 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Family History Positive | Family History Negative
Number analyzed (Participants) | 65 | 115
seconds
  Placebo: number analyzed (Participants) | 61 | 112
  Placebo | 75.27 (17.06) | 70.17 (12.03)
  Alcohol 40mg%: number analyzed (Participants) | 58 | 109
  Alcohol 40mg% | 75.19 (15.99) | 72.76 (14.29)
  Alcohol 100mg%: number analyzed (Participants) | 60 | 110
  Alcohol 100mg% | 85.86 (16.93) | 83.85 (16.48)

ADVERSE EVENTS:
Arm/Group | Family History Positive | Family History Negative
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/115
Other Adverse Events (participants affected / at risk) | 1/65 | 0/115
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Family History Positive (N=65) | Family History Negative (N=115)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes